CLINICAL TRIAL: NCT00280228
Title: Home-based Behavioral Therapy (HBT): Psychosocial Intervention Project for Early Adolescents With Pre- or Early Substance Use Disorder: Phase II
Brief Title: Home Based Treatment for Drug Use in Early Adolescents
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Oscar G. Bukstein, M.D., M.P.H., University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DA016631; 5R21DA016631 (NIH)
Record Dates: First submitted 2006-01-18; First posted 2006-01-20 (Estimated); Last update posted 2011-05-26 (Estimated); Status verified 2011-05

CONDITIONS: Attention Deficit Hyperactivity Disorder; Oppositional Defiant Disorder; Conduct Disorder; Substance Abuse
Keywords: ADHD; Oppositional Defiant Disorder; Conduct Disorder; Substance Use; Drug and Alcohol Use
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Oppositional Defiant Disorder; Conduct Disorder; Substance-Related Disorders; Alcohol Drinking | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Home Based Treatment
  Interventions: Behavioral: Adolescent Skills Parent Management Parent-Adol Negotiation
- 2 (Active Comparator): Treatment as Usual
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: Adolescent Skills Parent Management Parent-Adol Negotiation — Acute treatment for 12 weeks followed by three monthly booster sessions.
  Arms: 1
Behavioral: Treatment as Usual — Standard outpatient treatment for behavioral problems and substance use
  Arms: 2

SUMMARY:
This study will compare two programs to see if they are helpful in preventing the use of substances in adolescents with attention deficit-hyperactivity disorder (ADHD), oppositional defiant disorder (ODD), or conduct disorder (CD). One of the programs involves working with adolescents and their parent(s) in their home. The other program involves working with adolescents and their parent(s) in an office setting.

DETAILED DESCRIPTION:
In this study phase, 36 patients with a disruptive behavior disorder (DBD - i.e., attention deficit-hyperactivity disorder, oppositional defiant disorder, conduct disorder) and use or abuse of one or more substances will be randomly assigned to treatment using either a standard treatment for DBDs in this age group or the newly developed HBT treatment. Treatment outcomes for the 24 patients assigned to receive HBT will then be compared to outcomes for the 12 patients assigned to receive standard DBD treatment.

Specific aims of Phase II include:

1. finalizing the HBT treatment manual and measures of treatment fidelity, therapist competence, and treatment satisfaction;
2. generating estimates of treatment effect sizes for substance use, disruptive behavior, and functional status outcomes, as pilot data for a larger efficacy study, and
3. comparing treatment satisfaction for the two treatment groups.

We hypothesize that HBT will lead to significantly lower rates of disruptive behaviors, substance use, and SUDs than with standard treatment, as well as greater concomitant improvements in impairment.

ELIGIBILITY:
Inclusion Criteria:

* Study participants (subjects and parents) must provide written consent and verbal assent
* Adolescents aged 11 through 14 of any race or ethnic background,
* A DSM-IV disruptive behavior disorder diagnosis (either CD, ODD, ADHD or disruptive behavior disorder not otherwise specified [DBD NOS]),
* Adolescents who are either using one or more substances regularly (2 or more times a month for 3 consecutive months), and
* Acceptable insurance coverage (i.e., participant has insurance that is accepted by the University of Pittsburgh Medical Center [UPMC] in the event that they are randomly assigned to the treatment-as-usual [TAU] group).

Exclusion Criteria:

* Full scale IQ below 80;
* History of pervasive developmental disorder, schizophrenia or other psychotic disorders, organic mental disorders or eating disorders,
* Diagnosis of bipolar disorder,
* Recent treatment for substance problems, and/or
* Daily use of "hard" street drugs (i.e., cocaine, methamphetamine, heroin, inhalants).

Ages: 11 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Estimated)
Dates: Start 2006-01; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Rates of substance use and disruptive behaviors | immediately following acute 12 week treatment, at the end of 3 month followup, and at one year follow up

CONTACTS AND LOCATIONS:
Overall Officials: Oscar G Bukstein, M.D., M.P.H., Principal Investigator — University of Pittsburgh
Locations (1):
- Youth and Family Research Program, Pittsburgh, Pennsylvania, United States